CLINICAL TRIAL: NCT06317116
Title: Investigation of the Relationship Between Core Muscle Functions and Lower Urinary System Symptoms in Children
Brief Title: Examining the Relationship Between Core Muscles and Bladder Issues in Children
Status: Enrolling by invitation | Type: Observational
Sponsor: Izmir Bakircay University (Other)
Collaborators: Dokuz Eylul University (Other); Ege University Medical School (Other); The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Büşra PALAZ, Research Assistant, Izmir Bakircay University
Other Study IDs: 2023/09-14
Record Dates: First submitted 2024-03-11; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Lower Urinary Tract Symptoms; Skeletal Muscle
Keywords: lower urinary tract symptoms; children; physical therapy; core muscles
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about functional bladder problems in children. The main questions it aims to answer are:

* Does bladder symptoms in children have an effect on core muscles?
* How do core muscles change based on an increase or decrease in these symptoms?

DETAILED DESCRIPTION:
The study will be a novel investigation that elucidates the current state by comparing core muscle function outcomes with the type and severity of symptoms in children with lower urinary tract symptoms. It will shed light on the necessity of evaluating not only electromyographic activity during urination but also the overall function of core muscles in children with lower urinary tract symptoms. Additionally, identifying core muscle dysfunctions in children with lower urinary tract symptoms will provide a new perspective in treatment. Consequently, the project will not only contribute to the literature but also serve as a pioneering study that draws attention to the necessity of physical therapy consultation and a multidisciplinary approach in clinical assessment and treatment processes for pediatric urologists. The comprehensive and objective project aims to conduct a reference study on the subject, and the project results will lay the foundation for the development of prevention and improvement strategies. Data will be collected using non-invasive transabdominal ultrasound and surface electromyography to evaluate core muscle functions, and symptom questionnaires. The relationship between core muscle functions and lower urinary tract symptoms in children will be examined. Research Questions: Does lower urinary tract symptoms have an impact on core muscle functions in children? How do core muscle functions change according to an increase or decrease in these symptoms? The study is a cross-sectional research.

ELIGIBILITY:
Inclusion Criteria:

* To have a diagnosis of lower urinary tract symptoms according to the International Children's Continence Society (ICCS) diagnostic criteria,
* To have a normal neurological examination,
* Not to have received pelvic floor rehabilitation in the last 6 months,
* To be between the ages of 6 and 18.

Exclusion Criteria:

* To have structural (anatomical) problems in the urinary system such as ectopic ureter, urethral valve issues,
* To have congenital and/or spinal cord injury, acquired neurogenic problems such as spinal dysraphism, pelvic trauma,
* To have active febrile illness or urinary tract infection, or any biomechanical problem such as congenital thoracic deformities that may hinder or affect the evaluation,
* To have cognitive or mental impairment in the child and/or parent.

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients referred to the Pediatric Urology Clinic at Ege University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2024-09-29 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Dysfunctional Voiding and Incontinence Scoring System (DVAISS) | At the time of the initial physiotherapist examination
  DVAISS was developed to evaluate the severity of dysfunctional voiding and incontinence symptoms by Akbal et al. DVAISS consists of 14 questions examining daytime and nighttime symptoms, bladder and bowel habits, and quality of life. DVAISS score is based on the estimated odds ratio for each question between participants and controls. If the estimated odds ratio of the question is between 2 and 10, one point is given and if the estimated odds ratio is greater than 50, five points are given. The total score varies between 0 and 35. The increase in the total score indicates that the severity of the symptoms increases. A score of 8.5 or higher on the scale indicates the presence of bladder and bowel dysfunction. The Cronbach Alpha value of the scale was determined as 0.50.
Bladder and Bowel Dysfunction Questionnaire (BBDQ) | At the time of the initial physiotherapist examination
  BBDQ was developed to evaluate symptoms of bladder and bowel dysfunction by Afshar et al. The Turkish validity and reliability was conducted by Kaya Narter et al. BBDQ includes 13 questions about bladder and bowel symptoms such as incontinence, voiding, enuresis, dysuria, and constipation. Each question is scored on a 5-point Likert scale ranging from zero to four points. The total score varies between 0 and 52. As the total score increases, symptom severity worsens. A score of 11 points or above is considered bladder and bowel dysfunction. Cronbach Alpha value of the scale was found to be 0.727.
Childhood Bladder and Bowel Dysfunction Questionnaire (CBBDQ) | At the time of the initial physiotherapist examination
  CBBDQ consists of a total of 18 questions that assess bladder and bowel symptoms in children. CBBDQ has two subdimensions: Bladder Symptoms Scale (10 questions) and Bowel Symptoms Scale (8 questions). Considering the presence of children's symptoms in the last month, CBBDQ is filled out by parents on a 5-point Likert scale ranging from zero (no symptoms) to four points (symptoms occur almost every day). The total score from the scale varies between 0 and 72. As the total score increases, symptoms worsen. The Turkish validity and reliability of the scale was conducted by Aydin et al. Cronbach Alpha values were determined as 0.74 and 0.71 for bladder and bowel subdimensions, respectively.
Bladder Diary | two days
  The bladder diary is a simple and non-invasive method that objectively assesses bladder habits. The bladder diary is used to record the type and amount of consumed fluid over 48 hours, the amount and duration of urination, urgency, urinary frequency, and the amount and time of urinary incontinence. The bladder diary is desirable to record for two consecutive days. The amount of consumed fluid and the urination is expressed in milliliters (ml), and the duration of urination is expressed in seconds (sec).
Bowel Diary | seven days
  The ICCS recommends the use of a seven-day bowel diary in children with lower urinary tract symptoms due to the close relationship between bladder and bowel function. The bowel diary questions the defecation frequency, pain during defecation, urgency, stool type, and the presence of fecal incontinence. The Bristol Stool Scale is used for stool type. The bowel diary consists of seven pictures and stool form descriptors and allows children to express participants' bowel movement intensity.

SECONDARY OUTCOMES:
Superficial Electromyography (EMG) | At the time of the initial physiotherapist examination
  A NeuroTrac MyoPlus 4 PRO (Verity Medical LTD., UK) type EMG device will be used in the study. Bioelectrical activities of the muscles (pelvic floor muscles, abdominal muscles, diaphragm, multifidus) will be recorded with disposable 3.2 x 3.2 cm superficial electrodes. To reduce skin impedance, the skin area will be cleaned with an alcohol swab. Active electrodes will be placed on the right side of the body, parallel to the muscle fibers, according to the reference points. The reference electrode will be placed on the anterior superior iliac spine. Measurements will be performed during five seconds of maximal voluntary contraction ('work' phase EMG activity) and five seconds of relaxation ('rest' phase EMG activity) of the pelvic floor muscles. Measurements will be repeated for three times. The graphic and numerical data provided by the device will be recorded in the evaluation form.
Ultrasonography (USG) | At the time of the initial physiotherapist examination
  Pelvic floor displacement, endurance, phasic contraction and coordination, bladder volume, bladder wall thickness and post voiding residue, abdominal muscles and multifidus thicknesses, diaphragmatic displacement and thickness will be measured. A transabdominal diagnostic USG device (Sonospace SSI-600) with a low frequency (2-5 MHz) curvilinear transducer will be used. Muscle thickness and distance measurements will be made during frozen imaging. Muscle thickness will be measured between the upper border of the muscle fascia, which appears as a white line, and the end point of the lower border. Measurements will be taken at the expiration and during a five-second pelvic floor muscle contraction. Both measurement results will be recorded in millimeters. All measurements will be repeated three times and the average values will be noted on the evaluation form.

CONTACTS AND LOCATIONS:
Overall Officials: Özge Çeliker Tosun, Study Director — Dokuz Eylul University; Büşra Palaz, Principal Investigator — Izmir Bakircay University; İbrahim Ulman, Principal Investigator — Ege University; Ali Tekin, Principal Investigator — Ege University; Sibel Tiryaki Birol, Principal Investigator — Ege University; Nuray Elibol, Principal Investigator — Ege University; Barış Yücel, Principal Investigator — Ege University; Ezgi Altun Tanıl, Principal Investigator — Ege University
Locations (1):
- Ege University Hospital Pediatric Urology Outpatient Clinic, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No